CLINICAL TRIAL: NCT02109146
Title: A Randomized, Open-label, Phase 3 Trial Evaluating Adjuvant Transarterial Chemoembolization for TNM Stage I and II Hepatocellular Carcinoma Recurrence After Curative Resection
Brief Title: Postoperative TACE(Transhepatic Arterial Chemotherapy And Embolization) for Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-103
Record Dates: First submitted 2014-03-26; First posted 2014-04-09 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Hepatocellular Carcinoma; Transcatheter Arterial Chemoembolization
Keywords: TACE; Postoperation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Observation

STUDY DESIGN:
Intervention Model Description: After confirming eligibility by the investigators, patients without residual tumors on the CT/MRI were consented and randomly assigned in a 1:1 ratio into the adjuvant TACE group or the observation group. Allocation of treatment group was done with a computer-generated random number list.

ARMS (2):
- Adjuvant TACE (Experimental): Patients receive adjuvant Transcatheter Arterial Chemoembolization (TACE) following curative resection of HCC.
  Interventions: Drug: Prophylactic Transcatheter Arterial Chemoembolization
- Observation (Active Comparator): Patients do not receive TACE or any other adjuvant therapy following curative resection of HCC.
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Prophylactic Transcatheter Arterial Chemoembolization — Participants enrolled in the adjuvant TACE group received one to two cycles of TACE with an interval of 4~6 weeks, and the first TACE was given within 1 week after randomization.
  Arms: Adjuvant TACE
Other: Observation — Participants enrolled in the observation group were subjected to active surveillance without any adjuvant treatment.
  Arms: Observation

SUMMARY:
1. Hepatocellular carcinoma (HCC) is the most common primary malignancy of liver, representing the third leading cause of cancer-related death worldwide.
2. Its overall dismal prognosis is a result of high incidence rates of metastasis and postoperative recurrence, in particular the intrahepatic recurrence.
3. TACE is the most widely used primary treatment for unresectable HCC. It was also used as the optional treatment for relapsed disease. However, the efficacy of TACE used as adjuvant therapy following hepatectomy remains controversial.

DETAILED DESCRIPTION:
Eligible patients were between 18 and 75 years of age with histologically proven T1 or T2 HCC (according to the AJCC TNM Classification of HCC, 7th); an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; Child-Pugh class A or B; no history of neoadjuvant therapy; no lymph node or distant metastasis; no intrahepatic or extrahepatic recurrence at radiological follow-up (4-6 weeks after surgery); adequate bone marrow, hepatic, and renal function according to laboratory test results. Patients were excluded if they had undergone margin-positive resections or resection of recurrence HCC; had lymph node or distal metastases; underwent concomitant ablation or radiation during surgery; were subjected to severe postoperative complications; had serious co-morbidities; had known allergy to iodine and drugs used in TACE; or if an investigator judged participation to be incompatible with the safety of the study. This clinical trial was done in accordance with the Declaration of Helsinki and local laws. All participants provided written informed consent. The study protocol was approved by the institutional Medical Ethics Review Committee.

Participants enrolled in the adjuvant TACE group received one to two cycles of TACE with an interval of 4~6 weeks, and the first TACE was given within 1 week after randomization. Participants enrolled in the observation group were subjected to active surveillance without any adjuvant treatment. The TACE procedure was performed as follows. Briefly, a 4F or 5F catheter was introduced into the abdominal aorta through the superficial femoral artery according to the Seldinger technique. Angiography of the celiac and superior mesenteric arteries was performed to show the hepatic arterial supply. Then the left and right hepatic arteries were accessed by a microcatheter and intraarterial epirubicin (40 mg) and oxaliplatin (150 mg) in a mixture of lipiodol (3～5 mL) were injected. The follow-up interval was 3 months in the first two years postoperatively and 6 months thereafter. During each follow-up visit, blood tests including complete blood count, serum level of alpha-fetoprotein (AFP), and liver function tests were examined. During follow-up, contrast-enhanced abdominal CT or MRI scans were first performed at 3 months after operation and then every 6 months, with liver ultrasonography performed 3 months after every CT/MRI scan thereafter. Chest CT was performed at 1-year intervals. All participants with tumor recurrence were treated according to the decision made by a multidisciplinary board.

The primary endpoint was RFS, defined as the time from randomization to the first documented HCC recurrence by independent radiological assessment or death due to any cause, whichever occurred first. Secondary endpoints were OS (defined as the time from randomization to death due to any cause), RFS rate, and safety. Patients who were recurrence-free or alive at the point of final analysis were censored at the date of the last follow-up.

Intrahepatic recurrence was defined according to the non-invasive criteria of the European Association for the Study of the Liver (EASL) guideline. Newly-onset intrahepatic nodules with the longest diameter ≥ 1cm and a typical hallmark of HCC on contrast-enhanced CT/MRI imaging (hypervascular in the arterial phase with washout in the portal venous or delayed phase) were diagnosed as HCC recurrence. Lesions ≥ 1cm without a typical vascular pattern could also be diagnosed as HCC recurrence by evidence of a fast growth pattern as showed in subsequent scans and were independently reviewed by two radiologists. Extrahepatic recurrence was defined as per Response Evaluation Criteria in Solid Tumors. The safety of adjuvant TACE was assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of HCC (AJCC stage I or II)
* Without recurrence in 1 month postoperation
* Must be tolerant to TACE

Exclusion Criteria:

* With intrahepatic recurrence postoperation
* Insufficient liver function
* Stage III or IV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2023-05-13 (Actual); Study Completion 2023-05-13 (Actual)

PRIMARY OUTCOMES:
RFS(Recurrence free survival) | the time from randomization to the first documented HCC recurrence by independent radiological assessment or death due to any cause, whichever occurred first，assessed up to 120 months
  defined as the time from randomization to the first documented HCC recurrence by independent radiological assessment or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
OS (overall survival) | defined as the time from randomization to death due to any cause, assessed up to 120 months
  defined as the time from randomization to death due to any cause
RFS rate | the time from randomization to the first documented HCC recurrence by independent radiological assessment or death due to any cause, whichever occurred first，assessed up to 120 months
  defined as the time from randomization to the first documented HCC recurrence by independent radiological assessment or death due to any cause, whichever occurred first.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 24 weeks
  any adverse events recorded after TACE

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, M.D Ph.D, Study Chair — Zhejiang University
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China